CLINICAL TRIAL: NCT05118711
Title: COVID-19 Severity, Long-term Consequences for Exercise Capacity and Link to Associated Mechanisms
Brief Title: Sequelae of COVID-19 With Focus on Exercise Capacity and Underlying Mechanisms
Acronym: COR-PHYS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Arno Schmidt-Trucksäss (Other)
Responsible Party: Sponsor-Investigator, Arno Schmidt-Trucksäss, Sponsor-Investigator and Head of Rehabilitative and Regenerative Sports Medicine, Department of Sport, Exercise and Health, University of Basel
Organization: University of Basel (Other)
Other Study IDs: EKNZ 2021-01039
Record Dates: First submitted 2021-11-08; First posted 2021-11-12 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Patients Post-COVID-19; Controls
Keywords: SARS-CoV-2; Coronavirus; Sequelae; Exercise intolerance; Cardiopulmonary exercise testing
MeSH Terms: conditions — Coronavirus Infections | interventions — Cardiorespiratory Fitness; Respiration; Blood Specimen Collection; Exercise; Body Composition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples (total volume 36 mL) will be collected by venipuncture of the cubital fossa, are subsequently centrifuged and the plasma aliquots are frozen at -80°C.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 (18 months post-infection): Individuals with a positive Severe Acute Respiratory Syndrome-Coronavirus 2 (SARS-CoV-2) antigen-/polymerase chain reaction (PCR) test within the last 18 months that required hospitalisation. Symptoms typically worsened within a period of 5 to 10 days leading to e.g., prolonged fever, feeling of sickness and/or shortness of breath. This also includes individuals hospitalised in an intensive care ward. Individuals need to be hospitalised due to COVID-19 and not only with COVID-19.
  Interventions: Diagnostic Test: Cardiorespiratory fitness; Diagnostic Test: Lung function; Diagnostic Test: Muscular strength and balance tests; Diagnostic Test: Micro- and macrovascular endothelial function and cardiac function; Diagnostic Test: Blood sampling and analysis; Diagnostic Test: Physical activity; Diagnostic Test: Questionnaires; Diagnostic Test: Body composition
- Control group: Age-, sex-, and comorbidity-matched (frequency matching), fully vaccinated individuals with no history of symptomatic SARS-CoV-2 infection.
  Interventions: Diagnostic Test: Cardiorespiratory fitness; Diagnostic Test: Lung function; Diagnostic Test: Muscular strength and balance tests; Diagnostic Test: Micro- and macrovascular endothelial function and cardiac function; Diagnostic Test: Blood sampling and analysis; Diagnostic Test: Physical activity; Diagnostic Test: Questionnaires; Diagnostic Test: Body composition

INTERVENTIONS:
Diagnostic Test: Cardiorespiratory fitness — Cardiopulmonary exercise testing
Diagnostic Test: Lung function — Body plethysmography
Diagnostic Test: Muscular strength and balance tests — Handgrip strength test, mid-thigh pull test and standing balance test in static tandem stance
Diagnostic Test: Micro- and macrovascular endothelial function and cardiac function — Measurement of flow-mediated dilation, static and dynamic retinal vessel analysis, echocardiography
Diagnostic Test: Blood sampling and analysis — Blood sampling by venepuncture
Diagnostic Test: Physical activity — Physical activity surveillance using accelerometers
Diagnostic Test: Questionnaires — Global physical activity questionnaire (GPAQ), short-form 8 health survey (SF-8), barriers to physical activity, fatigue assessment scale (FAS), modified medical research council dyspnea scale (mMRC), depression, anxiety, and stress scale (DASS21), post-COVID-19 syndrome symptoms
Diagnostic Test: Body composition — Dual-energy x-ray absorptiometry (DXA)

SUMMARY:
The project is designed as a cross-sectional study and aims to examine long-term consequences of coronavirus disease 2019 (COVID-19) for selected bio-behavioural parameters while taking the disease course severity into account.

ELIGIBILITY:
Inclusion Criteria:

* tested positive for SARS-CoV-2 using antigen- or PCR tests within the last 18 months
* previous hospitalisation due to COVID-19
* fully vaccinated (only for controls)

Exclusion Criteria:

* inability to follow the study procedures (e.g. due to language barriers, psychological disorders, dementia, etc.),
* known pregnancy or lactating women,
* presence of any contraindications for exercising until maximum exhaustion, including insufficient blood pressure control (systolic >170 mmHg, diastolic >100 mmHg), ongoing cancer treatment, unstable angina pectoris, uncontrolled bradyarrhythmia or tachyarrhythmia, severe uncorrected valvular heart disease, clinically relevant acute infection, any form of musculoskeletal injury,
* participating in any interventional clinical trial within the last four weeks,
* previous participation in the current study
* history of symptomatic COVID-19 (only for controls)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Previously hospitalised patients recovering from COVID-19 and fully vaccinated controls with no history of symptomatic COVID-19.
  Recruitment of patients will be done via the University Hospital of Basel, Switzerland, the Clinic Barmelweid, Barmelweid, Switzerland, and Cantonal Hospital Olten, Olten, Switzerland. Participants for the control group will be recruited prospectively through unaddressed letters distributed in the Basel-Stadt area, newspaper, internet-based media, and word-of-mouth. Recruitment will continue until the number of valid datasets corresponds to the calculated sample size.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory fitness (as % of predicted V̇O2max) | 1.5 hours after inclusion in study
  Measured during cardiopulmonary exercise testing on a cycle ergometer.

SECONDARY OUTCOMES:
Forced expiratory volume in 1 s (as % of predicted) | 1.5 hours after inclusion in study
  Measured during bodyplethysmography.
Forced vital capacity (as % of predicted) | 1.5 hours after inclusion in study
  Measured during bodyplethysmography.
Total lung capacity (as % of predicted) | 1.5 hours after inclusion in study
  Measured during bodyplethysmography.
Diffusion capacity of the lungs (as % of predicted) | 1.5 hours after inclusion in study
  Measured during bodyplethysmography.
Muscle oxygenation at peak exercise (in %) | 1.5 hours after inclusion in study
  Measured using near-infrared spectroscopy during cardiopulmonary exercise testing on a cycle ergometer.
Cardiac output at peak exercise (in mL) | 1.5 hours after inclusion in study
  Measured non-invasive using the PhysioFlow device during cardiopulmonary exercise testing on a cycle ergometer.
Handgrip strength (in N) | 1 hour after inclusion in study
  Measured by a handheld dynamometer.
Handgrip rate of force development (in N/s) | 1 hour after inclusion in study
  Measured by a handheld dynamometer.
Macrovascular flow-mediated dilation at rest (in %) | 0.5 hours after inclusion in study
  Measured by ultrasound.
Microvascular flow-mediated dilation at rest (in %) | 2 to 14 days after inclusion in study
  Measured by retinal vessel analysis.
Fatigue Assessment Scale (FAS) score | 2 to 14 days after inclusion in study
  Scores range from 5 to 50 with higher scores indicating more severe fatigue.
Score of depression, anxiety, and stress questionnaire (DASS21) | 2 to 14 days after inclusion in study
  Scores range from 0 to 63 with higher scores indicating worse mental health.
Health distance | Calculated during statistical analysis
  The statistical (Mahalanobis) distance (health distance) is a composite measure of various health biomarkers
Cerebral oxygenation at peak exercise (in %) | 1.5 hours after inclusion in study
  Measured using functional near-infrared spectroscopy during cardiopulmonary exercise testing on a cycle ergometer.

CONTACTS AND LOCATIONS:
Overall Officials: Arno Schmidt-Trucksäss, Prof., Principal Investigator — Department of Sport, Exercise and Health, University of Basel, Basel, Switzerland
Locations (1):
- Division of Sports and Exercise Medicine, Department of Sport, Exercise and Health, University of Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No